CLINICAL TRIAL: NCT02094729
Title: A Randomized, Double-blind, Placebo-controlled Study to Assess Safety, Tolerability, Pharmacokinetics, Immunogenicity, and Pharmacodynamic Response of Repeated Intravenous Infusions of BAN2401 in Subjects With Mild Cognitive Impairment Due to Alzheimer's Disease and Mild Alzheimer's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BAN2401-J081-104
Record Dates: First submitted 2014-01-09; First posted 2014-03-24 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-06

CONDITIONS: Alzheimer's Disease
Keywords: mild cognitive impairment; Alzheimer's disease
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction | interventions — lecanemab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- BAN2401 2.5 mg/kg (Experimental): Cohorts 1: Intravenous infusions of 2.5 mg/kg BAN2401
  Interventions: Drug: BAN2401 2.5 mg/kg
- BAN2401 5 mg/kg (Experimental): Cohorts 2: Intravenous infusions of 5 mg/kg BAN2401
  Interventions: Drug: BAN2401 5 mg/kg
- BAN2401 10 mg/kg (Experimental): Cohorts 3: Intravenous infusions of 10 mg/kg BAN2401
  Interventions: Drug: BAN2401 10 mg/kg
- Placebo (Placebo Comparator): Intravenous infusions of placebo for 60 +/- 10 minutes.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BAN2401 2.5 mg/kg — Cohorts 1: Intravenous infusions of 2.5 mg/kg BAN2401 for 60 +/- 10 minutes.
  Arms: BAN2401 2.5 mg/kg
Drug: BAN2401 5 mg/kg — Cohorts 2: Intravenous infusions of 5 mg/kg BAN2401 for 60 +/- 10 minutes.
  Arms: BAN2401 5 mg/kg
Drug: BAN2401 10 mg/kg — Cohorts 3: Intravenous infusions of 10 mg/kg BAN2401 for 60 +/- 10 minutes
  Arms: BAN2401 10 mg/kg
Drug: Placebo — Intravenous infusions of placebo for 60 +/- 10 minutes.
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the safety, tolerability, pharmacokinetics, immunogenicity, and pharmacodynamic response of repeated intravenous infusions of BAN2401 in subjects with mild cognitive impairment (MCI) due to Alzheimer's disease (AD) and mild Alzheimer's disease.

DETAILED DESCRIPTION:
This is a multicenter, randomized, placebo-controlled, double-blind, multiple ascending dose study in a total of 24 subjects (8 subjects per cohort) with MCI due to AD and mild AD. The study consists of three cohorts to evaluate the safety, tolerability and PK of BAN2401 at three dose levels (2.5, 5, and 10 mg/kg). Each cohort consists of Screening Period before randomization, Treatment Period from randomization to last dose, and Follow-up Period after last dose. Cohorts 1, 2, and 3 will receive 2.5 mg/kg, 5 mg/kg, and 10 mg/kg of BAN2401, respectively.

ELIGIBILITY:
Inclusion Criteria

MCI due to AD

1. Subjects who have clinical and cognitive symptoms consistent with the National Institute on Aging-Alzheimer's Association (NIA-AA) core criteria for MCI
2. Subjects who have a Clinical Dementia Rating (CDR) of 0.5 and a memory box score of 0.5 or greater at Screening
3. Subjects who report a history of subjective memory decline with slow progression at least 1 year before Screening, or subjects whose information provider or attending physician reports a history of memory decline with slow progression at least 1 year before Screening
4. Subjects with objective impairment in episodic memory as indicated by 1-1.5 standard deviations below age-adjusted mean in the Wechsler Memory Scale-Revised (WMS-R) logical memory II (delayed recall) at Screening:

   * less than or equal to 15 for age 50 to 64 years
   * less than or equal to 12 for age 65 to 69 years
   * less than or equal to 11 for age 70 to 74 years
   * less than or equal to 9 for age 75 to 79 years
   * less than or equal to 7 for age 80 to 90 years

   Mild AD
5. Subjects who meet the NIA-AA core clinical criteria for probable AD
6. Subjects who have a CDR of 0.5 or 1.0 and a memory box score of 0.5 or greater at Screening

   All subjects
7. Male or female subjects aged between 50 and 90 years, inclusive, at obtaining informed consent
8. Subjects who have an Mini Mental State Examination (MMSE) score greater than or equal to 22 and less than or equal to 30 at Screening
9. Body Mass Index (BMI) less than 35 kg/m2 at Screening
10. Females must not be pregnant or lactating, and specified contraceptive precautions must be followed
11. Subjects must have identified caregivers/informants
12. Must have an informant or a caregiver who will provide written informed consent voluntarily and is able to spend 3 days a week with the subject (4 hours per day), and is able to support the subject during the study period by providing necessary patient information, assisting treatment compliance, and accompanying the subject to all scheduled visits (if needed) throughout the study.
13. Provide voluntary written informed consent (obtaining as much as possible from subjects, but mandatory from their legal guardians).
14. Willing and able to comply with all aspects of the protocol.

Exclusion Criteria

1. Any neurological condition that may affect cognitive impairment
2. History of transient ischemic attacks (TIA), stroke, or seizures within 12 months of Screening
3. Any psychiatric diagnosis or symptoms (e.g., hallucinations, major depression, or delusions) that could interfere with study procedures in the subject
4. Any medical devices contraindicated for MRI scanning (e.g., cardiac pacemaker/defibrillator, ferromagnetic metal implants, any devices other than those approved as safe for use in MRI scanners)
5. Evidence of infection, tumor, stroke or other clinically significant lesions that could indicate a dementia diagnosis other than AD on brain MRI at Screening
6. Evidence of other clinically significant lesions that could indicate a dementia diagnosis other than AD on brain MRI at Screening, or other significant pathological findings on brain MRI at Screening
7. A prolonged QT interval (QTcF greater than or equal to 450 ms) as demonstrated by a repeated ECG at Screening
8. Any other clinically significant conditions (e.g., cardiac, respiratory, gastrointestinal, renal disease) that in the opinion of the investigator(s) could affect the subject's safety or interfere with the study assessments
9. Severe visual or hearing impairment that would prevent the subject from performing psychometric tests accurately.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2013-09; Primary Completion 2015-03 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | Up to 14 weeks
  Safety assessment variables will include all adverse events (AEs) including serious and non-serious AEs; laboratory parameters (hematology, blood chemistry, and urinalysis); vital signs; electrocardiograms; and physical examination; as well as a risk of suicide using C-SSRS and brain MRI.

SECONDARY OUTCOMES:
Pharmacokinetics of BAN2401: Maximum Concentration (Cmax) | Up to 14 weeks
  Cmax after single and repeated administrations based on non-compartmental analysis.
Pharmacokinetics of BAN2401: time attain to Cmax (tmax) | Up to 14 weeks
  tmax after single and repeated administrations based on non-compartmental analysis.
Pharmacokinetics of BAN2401: Area under the curve (AUC) | Up to 14 weeks
  AUC after single and repeated administrations based on non-compartmental analysis.
Pharmacokinetics of BAN2401: Drug Clearance (CL) | Up to 14 weeks
  CL after single and repeated administrations based on non-compartmental analysis.
Pharmacokinetics of BAN2401: apparent volume of distribution at steady state (Vss) | Up to 14 weeks
  Vss after single and repeated administrations based on non-compartmental analysis.
Investigation of the effect of repeated intravenous infusions of BAN2401 on the immunogenicity and CSF biomarkers | Up to 14 weeks
  Summary statistics (mean, standard deviation, median, minimum and maximum) will be calculated for each measurement of CSF concentrations of AB1-40, AB1-42, AB1-x, total tau and p-tau and their percent changes from baseline.
Investigation of the effect of apolipoprotein allele4 (ApoE4) on the safety, tolerability and pharmacodynamic (PD) response of repeated intravenous infusions of BAN2401 | Up to 14 weeks

CONTACTS AND LOCATIONS:
Locations (4):
- Japan (4):
  - Kobe, Hyōgo
  - Sendai, Miyagi
  - Kurashiki, Okayama-ken
  - Koto-ku, Tokyo